CLINICAL TRIAL: NCT00439049
Title: General Evaluation of Eligibility for Substance Abuse/Dependence Research
Brief Title: Substance Abuse Pre-Treatment Screening Study
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psy, Behavioral Science, The University of Texas Health Science Center, Houston
Other Study IDs: NIDA-09262-13; P50DA009262 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Cocaine Abuse; Cocaine Dependence; Opiate Dependence; Alcohol Dependence; Substance Abuse
Keywords: Substance Abuse; Treatment; Eligibility
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Alcoholism; Substance-Related Disorders | interventions — Modafinil; Dextroamphetamine; Levodopa; carbidopa, levodopa drug combination; Naltrexone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Cocaine Dependent Subjects
  Interventions: Drug: modafinil; Drug: d-amphetamine; Drug: L-Dopa; Drug: Naltrexone

INTERVENTIONS:
Drug: modafinil — 400 mg daily
  Other Names: Provigil
Drug: d-amphetamine — 60mg daily
  Other Names: Dexedrine
Drug: L-Dopa — 800/200mg daily
  Other Names: Sinemet
Drug: Naltrexone — 50mg daily
  Other Names: Revia

SUMMARY:
The overarching goal of this project is to have a consolidated consent and evaluation procedure that will lead potential subjects to the most appropriate clinical trial or human laboratory study (and its consent process) for their presenting concerns or interests. A second purpose is to have a consolidated intake data base on which secondary analyses can be conducted.

DETAILED DESCRIPTION:
Approximately 1500 candidates per year will respond to advertisements and will complete preliminary telephone screening without identifiers. Appropriate candidates will be given appointment times and on arrival will undergo the consent process for evaluation. A complete medical, social, psychiatric, and drug use history will be obtained. Subjects fulfilling general health inclusion requirements will then be offered an appropriate study for which the specific consent will be obtained. The evaluation period will be no more than one day with all results evaluated within the two following days. Acceptable candidates will then be invited to complete the study specific consent.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate in 3- to 6-month treatment program.
* At least 18 years of age.
* Seeking treatment for substances of abuse including (cocaine, opiates, and alcohol).
* Generally physically healthy.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Mandated by the courts/parole officers to attend treatment.
* Not seeking treatment for substances of abuse.
* Plans to move from the Houston area within the 3- to 6-month treatment period.
* Seeking treatment for a substance for which the Treatment Research Clinic (TRC) has no current trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cocaine Dependent Subjects
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2005-10; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Urine Toxicology | 6 weeks to 24 weeks

SECONDARY OUTCOMES:
Demographics | 6 weeks to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joy M. Schmitz, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Frederick G Moeller, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Angela L Stotts, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Medical School- Houston, Dept. of Psychiatry Mental Sciences Institute, Houston, Texas, United States